CLINICAL TRIAL: NCT01326715
Title: Manganese-Enhanced Magnetic Resonance Imaging in Healthy Volunteers and People With Multiple Sclerosis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 110116; 11-N-0116
Record Dates: First submitted 2011-03-30; First posted 2011-03-31 (Estimated); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Multiple Sclerosis
Keywords: Mangafodipir; Brain; MEMRI; Healthy Volunteer; Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — N,N'-bis(pyridoxal-5-phosphate)ethylenediamine-N,N'-diacetic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- mangafodipir (Active Comparator): see protocol
  Interventions: Drug: Mangafodipir (Teslascan)

INTERVENTIONS:
Drug: Mangafodipir (Teslascan) — gadolinium enhancement on contrast enhanced brain MRI.

SUMMARY:
Background:

- Contrast agents are drugs that make certain body areas or abnormalities show up better on imaging studies, such as magnetic resonance imaging (MRI) scans. Mangafodipir is an MRI contrast agent with manganese that has been approved for MRI scans of the liver and pancreas. Because contrast agents with manganese have also been shown to be useful in studying problems with the nervous system, researchers are interested in determining if mangafodipir may be used for MRI scans of the brain or eye, two areas that often experience problems caused by disorders that affect the nervous system, such as multiple sclerosis. However, more information is needed on whether mangafodipir will be useful for this purpose, or how best to use it in MRI scans of the eye and brain. To study mangafodipir more closely, researchers are interested in studying its use in both individuals with multiple sclerosis and healthy volunteers.

Background:

- Contrast agents are drugs that make certain body areas or abnormalities show up better on imaging studies, such as magnetic resonance imaging (MRI) scans. Mangafodipir is an MRI contrast agent with manganese that has been approved for MRI scans of the liver and pancreas. Because contrast agents with manganese have also been shown to be useful in studying problems with the nervous system, researchers are interested in determining if mangafodipir may be used for MRI scans of the brain or eye, two areas that often experience problems caused by disorders that affect the nervous system, such as multiple sclerosis. However, more information is needed on whether mangafodipir will be useful for this purpose, or how best to use it in MRI scans of the eye and brain. To study mangafodipir more closely, researchers are interested in studying its use in both individuals with multiple sclerosis and healthy volunteers.

Objectives:

- To evaluate the safety and effectiveness of mangafodipir in imaging studies of nerve disorders affecting the eye and brain.

Eligibility:

- Individuals between 18 and 70 years of age who either have been diagnosed with multiple sclerosis or are healthy volunteers.

Design:

* Participants will be screened with a physical examination, medical history, and blood tests.
* Participants will have up to 10 outpatient visits for screening and MRI scans over a period of up to 2 months. Participants will be divided into Eye and Brain groups, based on which area will be studied during the scans. (Participants who have available time may be eligible for study in both groups.)
* Participants will have an initial MRI scan as part of the screening process.
* At the first visit, participants will have a baseline MRI scan once before receiving mangafodipir.
* Participants will have up to five MRI scans, with the following procedures:
* Eye imaging group: MRI scans will be scheduled at specific times between 2 and 48 hours after receiving mangafodipir. Eye MRI participants will wear a dark contact lens and an eye patch for 30 minutes before receiving mangafodipir, and leave both on for up to 8 hours. The other eye will remain uncovered.
* Brain imaging group: MRI scans will be scheduled at specific times between 48 hours and 7 days after receiving mangafodipir.
* Participants will have a follow-up MRI scan 1 month after receiving mangafodipir. This scan is done to see how long mangafodipir may affect MRI images of the brain.

DETAILED DESCRIPTION:
Objective

The original goals of this pilot study were to assess whether: (1) manganese-enhanced magnetic resonance imaging (MEMRI) using mangafodipir trisodium, a contrast agent that enters the intracellular compartment, can detect multiple sclerosis-related tissue damage in the retina, optic nerve, and brain; and (2) the MRI effects of manganese are detectable in the basal ganglia one month following administration. With amendment F, the retina and optic nerve portions of the study have been eliminated, and we have modified our focus to examination of participants with multiple sclerosis and MRI evidence of abnormal permeability to gadolinium. In these individuals, mangafodipir may allow assessment of brain connectivity that is not possible to achieve with a gadolinium-based contrast agent, which remains in the extracellular space.

Study Population

Up to 15 healthy volunteers and up to 15 participants with multiple sclerosis.

Design

The first phase of the study involved healthy volunteers and focuses on optimizing our imaging protocol. The second phase studies participants with multiple sclerosis. With amendment F, the focus has shifted to evaluating participants with multiple sclerosis and evidence of gadolinium enhancement on contrast-enhanced brain MRI.

We have completed enrollment of 15 healthy volunteers. With Amendment G, we will remove references to the enrollment and screening procedures for healthy volunteers.

Outcome Measures

The primary outcome measure is T1-weighted signal intensity, measured: (1) in the retina, optic nerve, and brain at early time points after mangafodipir administration; and (2) in the basal ganglia, cerebral cortex, and whole brain one month following administration.

ELIGIBILITY:
* This study enrolls two cohorts:
* Up to 15 healthy volunteers
* Up to 15 MS patients

INCLUSION CRITERIA:

* Age 18 to 70 (inclusive)
* Able to give informed consent
* Able to comply with study procedures
* Diagnosis of multiple sclerosis according to the current McDonald Criteria
* Evidence of abnormal permeability of the brain or cerebrospinal fluid, based on a screening gadolinium-enhacned MRI scancan

EXCLUSION CRITERIA:

* Reported history of clinically significant medical disorders, such as liver or kidney disease, that could potentially increase the risk of CNS damage due to manganese exposure
* Uncontrolled hypertension, demonstrated by a blood pressure reading of >160/100 at screening on repeat exam
* Screening labs demonstrating any value for hepatic or biliary function out of the range of normal, to include AST, ALT, bilirubin, gammaGT, alkaline phosphatase; repeat value of the same test showing normal results will remove the exclusion
* For patients receiving ocular MRI, reported history of ocular disorders
* Previous or current alcohol and/or substance abuse
* Previous presumed occupational exposure to manganese (i.e., having worked in a mine, foundry, smelter, dry cell battery manufacturing facility, or agriculture)
* Medical contraindications for MRI (e.g., any non-organic implant or other device such as a cardiac pacemaker or infusion pump or other metallic implants, objects or body piercings that are not MRI-safe or that cannot be removed)
* Psychological contraindications for MRI (e.g., claustrophobia), to be assessed at the time the medical history is collected
* Pregnancy or current breastfeeding
* Allergy to manganese
* Reported history of impaired hearing, because people with impaired hearing are at increased risk of sound-induced damage from the MRI scanner
* Ongoing treatment with calcium-channel blockers
* Clinically significant iron-deficiency anemia

  * 5 contrast-enhancing lesion on screening MRI performed within one week of administration of mangafodipir

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2013-10-17 (Actual); Primary Completion 2019-09-18 (Actual); Study Completion 2022-09-13 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure is normalized T1-weighted signal intensity. | early time points after mangafodipir administration
  T1#weighted signal intensity, measured in selected brain structures at early time points after mangafodipir administration, as well as inthe basal ganglia, cerebral cortex, and whole brain one month following administration.

CONTACTS AND LOCATIONS:
Overall Officials: Daniel S Reich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- [Background] Andrews HE, Nichols PP, Bates D, Turnbull DM. Mitochondrial dysfunction plays a key role in progressive axonal loss in Multiple Sclerosis. Med Hypotheses. 2005;64(4):669-77. doi: 10.1016/j.mehy.2004.09.001. PMID 15694681
- [Background] Aoki I, Wu YJ, Silva AC, Lynch RM, Koretsky AP. In vivo detection of neuroarchitecture in the rodent brain using manganese-enhanced MRI. Neuroimage. 2004 Jul;22(3):1046-59. doi: 10.1016/j.neuroimage.2004.03.031. PMID 15219577
- [Background] Aschner M, Guilarte TR, Schneider JS, Zheng W. Manganese: recent advances in understanding its transport and neurotoxicity. Toxicol Appl Pharmacol. 2007 Jun 1;221(2):131-47. doi: 10.1016/j.taap.2007.03.001. Epub 2007 Mar 12. PMID 17466353
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2011-N-0116.html